CLINICAL TRIAL: NCT01842126
Title: Study of Safety, Tolerability, and Pharmacokinetics of BG00010 (Neublastin) Intravenous and Subcutaneous Single Ascending Doses in Healthy Volunteers, and Subcutaneous Multiple Ascending Doses in Subjects With Painful Lumbar Radiculopathy
Brief Title: Phase 1 Subcutaneous Single and Multiple Ascending Dose Study of BG00010 (Neublastin)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 103NS103; 2012-005224-15 (EudraCT Number)
Record Dates: First submitted 2013-04-25; First posted 2013-04-29 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-02

CONDITIONS: Painful Lumbar Radiculopathy; Healthy
Keywords: Sciatica
MeSH Terms: conditions — Sciatica | interventions — Nerve Growth Factor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Single Ascending Dose (SAD): BG00010 (Experimental): Up to five cohorts of healthy volunteers will receive a single dose of intravenous (IV) BG00010 followed by a single SC dose of BG00010 2 weeks apart.
  Interventions: Biological: BG00010 IV; Biological: BG00010 SC
- SAD: Placebo (Experimental): Up to five cohorts of healthy volunteers will receive a single IV dose of placebo followed by a single SC dose of placebo 2 weeks apart.
  Interventions: Drug: Placebo IV; Drug: Placebo SC
- Multiple Ascending Dose (MAD): BG00010 (Experimental): Up to 6 cohorts of participants with painful lumbar radiculopathy will receive 3 SC doses of BG00010.
  Interventions: Biological: BG00010 SC
- Multiple Ascending Dose (MAD): Placebo (Experimental): Up to 6 cohorts of participants with painful lumbar radiculopathy will receive 3 SC doses of placebo.
  Interventions: Drug: Placebo SC

INTERVENTIONS:
Biological: BG00010 IV — Ascending Doses intravenous (IV) of BG00010
  Other Names: Neublastin
  Arms: Single Ascending Dose (SAD): BG00010
Biological: BG00010 SC — Ascending Doses subcutaneous (SC) of BG00010
  Other Names: Neublastin
  Arms: Multiple Ascending Dose (MAD): BG00010; Single Ascending Dose (SAD): BG00010
Drug: Placebo IV — Ascending Doses intravenous (IV) of Placebo
  Arms: SAD: Placebo
Drug: Placebo SC — Ascending Doses subcutaneous (SC) of placebo
  Arms: Multiple Ascending Dose (MAD): Placebo; SAD: Placebo

SUMMARY:
The primary objective of the study is to evaluate the safety and tolerability of a range of single intravenous (IV) and subcutaneous (SC) doses of BG00010 in healthy volunteers, and a range of multiple SC doses of BG00010 in participants with painful lumbar radiculopathy. Secondary objectives of this study are to determine the single IV and SC dose pharmacokinetics (PK) profile of BG00010 in healthy volunteers including assessment of bioavailability by comparing SC exposure to IV exposure in each participant, to determine the multiple SC dose PK profiles of BG00010 in participants with painful lumbar radiculopathy, to assess the single IV and SC dose immunogenicity of BG00010 in healthy volunteers, to assess the multiple SC dose immunogenicity of BG00010 in participants with painful lumbar radiculopathy, and to assess the potential of BG00010 to reduce pain following multiple SC administrations in participants with painful lumbar radiculopathy.

ELIGIBILITY:
Key Inclusion Criteria: Part I and Part II

* Healthy Volunteers

Key Inclusion Criteria: Part III multiple ascending dose (MAD)

* Subjects must have a diagnosis of unilateral painful lumbar radiculopathy and painful lumbar radiculopathy symptoms must be present for 3 or more months prior to the Screening Visit.
* Subjects must rate their pain at ≥40 mm on the 100 mm visual analog scale (VAS) of the short form McGill pain questionnaire (SF-MPQ) at the Screening and Baseline Visits.

Key Inclusion Criteria for All Subjects for Part I, Part II, Part III:

* All male subjects and all female subjects of childbearing potential must practice effective contraception during the study and be willing and able to continue contraception for 3 months after their last dose of study treatment. -

Key Exclusion Criteria for All Subjects for Part I, Part II, Part III:

* History of or positive screening test for hepatitis C infection , hepatitis B infection, or positive for human immunodeficiency virus (HIV) antibody. Subjects who are hepatitis B surface antigen (HBsAg) negative and hepatitis B core antibody (HBcAb) positive are allowed to participate if they are positive for HBsAb immunoglobulin G
* History of malignancy or clinically relevant (as determined by the Investigator) allergies; cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic (not related to painful lumbar radiculopathy), dermatologic, rheumatic/joint, psychiatric, renal, and/or other major disease.
* Relevant history of illicit drug or alcohol abuse (as defined by the Investigator) within 1 year prior to the Screening Visit. -
* Female subjects who are pregnant or currently breastfeeding, or who have a positive pregnancy test result at the Screening or Baseline Visits.
* Previous administration of a neurotrophic factor, including BG00010.
* Participation in a study with another investigational drug or approved therapy for investigational use within the 3 months prior to the Baseline Visit, or current enrollment in any other study.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2013-04; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
The number of participants with Adverse Events (AEs)/Serious Adverse Events (SAEs) | Up to Day 75

SECONDARY OUTCOMES:
Maximum observed concentration (Cmax) of BG00010 | Pre-dose and up to 24 hours post-dose
Time to maximum serum concentration (Tmax) of BG00010 | Pre-dose and up to 24 hours post-dose
Half life (t1/2) of BG00010 | Pre-dose and up to 24 hours post-dose
Area under the serum concentration time curve (AUC) from zero to infinity AUC(0-∞) for BG00010 | Pre-dose and up to 24 hours post-dose
Subcutaneous (SC) bioavailability | Pre-dose and up to 24 hours post-dose
Number of participants with anti-BG00010 antibodies in serum | Up to Day 75
Pain as measured by an 11-point numeric rating scale (NRS) | Up to Day 75
  The Numeric Rating Scale (NRS-11) is an 11-point scale for patient self-reporting of pain. The scale ranges from 0 (no pain) to 10 (worst pain imaginable).
Pain as measured by short form McGill pain questionnaire (SF-MPQ) visual analog scale (VAS) | Up to Day 75
  A 10 cm visual analog scale ranging from 0 (no pain) to 10 (worst possible pain).

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Center for Human Drug Research, Leiden, Netherlands